CLINICAL TRIAL: NCT00689455
Title: Regional Observatory on Metabolic Syndrome in Italy- LAZIO
Brief Title: Regional Observatory on Metabolic Syndrome- LAZIO
Acronym: ORSA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Mario Mangrella MD Medical Manager, Cardiometabolic Team, AstraZeneca S.p.A.
Other Study IDs: NIS-CIT-DUM-2008/2
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Lipids; Waist Circumference
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Primary care population

SUMMARY:
The aim of the study, is to assess the prevalence of Metabolic Syndrome in Italy on a regional basis, defined according to NCEP/ATPIII Guidelines criteria.

ELIGIBILITY:
Inclusion Criteria:

* lipid profile in the last year
* Signed informed consent

Exclusion Criteria:

* Subjects with serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's successful participation in the study
* Pregnancy or breast feeding
* Subject who are unwilling or unable to provide the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1574 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of Metabolic Syndrome in Primary Care Population. | At Visit

SECONDARY OUTCOMES:
Concomitant presence of other CV risk factors. | At Visit

CONTACTS AND LOCATIONS:
Overall Officials: Volpe Massimo, MD, FACC, Study Chair — Cardiology Dept. Director, Sapienza University, Sant' Andrea Hospital, Rome
Locations (3):
- Italy (3):
  - Research Site, Rieti
  - Research Site, Rome
  - Research Site, Viterbo